CLINICAL TRIAL: NCT05253586
Title: A Single Blinded Randomised Controlled Trial Comparing the Ergonomics of Laparoscopic and Versius Robotic Assisted Abdominal Hernia Surgery
Brief Title: Versius or Laparoscopic Abdominal Hernia REpair
Acronym: VOLARE
Status: Withdrawn | Type: Observational
Why Stopped: PhD studentship research defined area changed.
Sponsor: Joanne Turner (Other Government)
Responsible Party: Sponsor-Investigator, Joanne Turner, Academic Research Coordinator, Milton Keynes University Hospital NHS Foundation Trust
Organization: Milton Keynes University Hospital NHS Foundation Trust (Other Government)
Other Study IDs: MKUH-RD-019
Record Dates: First submitted 2022-01-04; First posted 2022-02-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Hernia; Abdominal Surgery
Keywords: ergonomics; robotics; versius
MeSH Terms: conditions — Hernia, Abdominal | interventions — Laparoscopy; Robotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Laparoscopic Arm: This cohort of participants will have their procedure completed by a human surgeon.
  Interventions: Procedure: Laparoscopic
- Robotic Arm: This cohort of participants will have their procedure completed by the Versius Surgical Robotic System.
  Interventions: Procedure: Robotic

INTERVENTIONS:
Procedure: Laparoscopic — Surgeon
  Groups: Laparoscopic Arm
Procedure: Robotic — Versius system
  Groups: Robotic Arm

SUMMARY:
This trial will compare laparoscopic and robotic-assisted abdominal hernia repairs, using the Versius® system. We will initially aim to recruit 60 patients (20 patients in the laparoscopic arm and 40 in the robotic arm) in order to assess the ergonomic impact of each modality on the operating surgeon. This aims to provide in vivo information on whether robotic surgery provides any advantages to the operating surgeon. This trial will also be used to assess the feasibility of recruitment to a future larger study, and any data collected will be used as pilot data.

DETAILED DESCRIPTION:
This study has been designed to assess the ergonomics of Versius® assisted surgery in comparison with laparoscopic surgery in the management of abdominal hernias. The study will randomise 60 patients who require repair of an abdominal hernia and have been deemed suitable for a minimally invasive approach. Patients will be randomised to receive either laparoscopic or Versius® robotic assisted surgery but will be informed that it will be attempted via a minimally invasive approach that could include either of these two subtypes of minimally invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Need for abdominal hernia repair surgery

  * Incisional
  * Congenital
* Deemed suitable for minimally invasive surgery

Exclusion Criteria:

* Patients who are unable to consent
* Prisoners
* Patients in need of emergency surgery
* Patients with a hernial defect size of over 7cm

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pateints diagnosed with an abdominal hernia and are deemed suitable for minimally invasive surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
To compare the operating surgeon ergonomics (physical strain) of laparoscopic and Versius® robotic assisted surgery | Length of the procedure expected to be between 1-4 hours
  body position (physical strain) and cognitive workload (mental strain) assessed using the REBA score

SECONDARY OUTCOMES:
Measurement of the rate of participant recruitment | Through study completion, an average of 1 year.
  Measure the number of participants recruited over the length of time. The units of measurement will be presented on a scale of number of participants over a predetermined length of time.
Measurement of drop-out (withdrawal) rate of participants | Assessed from Day 1 (Randomisation) to date of withdrawal
  Measure the number of participants who withdrawal (drop out) from the trial. The units of measurement will be presented on a scale of numbers of withdrawals versus time.
Measurement of the unblinding rate of participants | Through study completion, an average of 1 year.
  Measure the number of participants where the treatment is unblinded during the trial. This is measured by the number of participants over the length of time who's treatment is unblinded.
Mental strain of surgeon | 30 minutes maximum completion time per surgeon
  To compare the operating surgeon mental strain of each approach using the NASA-Task Load Index score.
Health Economics | Procedure and recovery inpatient stay per participant expected to be between 1-3 days.
  Explore health economic aspects of each approach via calculation of the entire hospital episode and individual operation (including fixed costs and instrument costs) comparing the cost for cohort using the Versus Surgical Robot versus the human surgeon.
Communication | 1-4 hours expected for the duration of the procedure
  To compare differences in in-theatre communication assessed from audiovisual footage, using the Oxford NOTECHS II score.
Satisfaction with life scale | Assessed on Day 14
  Quality of life units completion of EQ-5D-5L questionnaire post operatively on day 14. Total scores used not sub scales to be reported.
Satisfaction with life scale | Assessed on Day 14
  Quality of life units completion of MFSI-SF questionnaires post operatively on day 14. Total scores used not sub scales to be reported.
Length of in-patient stay | Up to 4 weeks
  Measure of the time in days of each participant's hospital stay as an in-patient.
Pain Scores | Days 1, 2, 3, 14 and 28
  Using a uni-dimensional pain score measurement examining the change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Keeler, Principal Investigator — Consultant Colorectal Surgeon

IPD SHARING:
Plan to Share IPD: No